CLINICAL TRIAL: NCT05457023
Title: A Blood Biomarker for Sports-Related Brain Injury and Its Relationship With Omega-3 Status and Purposeful Soccer Heading in Free-Living Collegiate Women Soccer Players During and After a Competitive Season
Brief Title: Plasma Neurofilament Light and Its Relationship With Omega-3 Status and Soccer Heading in Women Soccer Players
Status: Completed | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Aaron Carbuhn, Assistant Professor, University of Kansas Medical Center
Other Study IDs: STUDY00148618
Record Dates: First submitted 2022-07-07; First posted 2022-07-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Brain Trauma
Keywords: Soccer, Heading, Omega-3, Neurofilament Light, Subconcussive, Women
MeSH Terms: conditions — Brain Injuries, Traumatic; Charcot-Marie-Tooth disease, Type 1F

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Collegiate Women Soccer Players: National Collegiate Athletic Association (NCAA) players.
  Interventions: Other: Plasma Neurofilament Light (NF-L); Other: Omega-3 Index; Other: HeadCount Questionnaire

INTERVENTIONS:
Other: Plasma Neurofilament Light (NF-L) — Plasma NF-L is a biomarker of axonal brain injury following sports-related head impacts.
Other: Omega-3 Index — Omega-3 Index is the omega-3 fatty acid content of eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) within the erythrocyte cell membrane. It is expressed as EPA+DHA as a percent of total identified fatty acids.
Other: HeadCount Questionnaire — HeadCount is a web-based, structured, self-administered questionnaire to assess longer-term heading exposure during competitive play and is administered bi-weekly.

SUMMARY:
The purpose of this study is to (1) assess how a competitive season of purposeful gameplay soccer heading in collegiate women soccer players is related to a blood biomarker for sports-related brain injury, plasma neurofilament light (NF-L), and (2) examine how a player's omega-3 status is related to plasma NF-L concentration changes during and after a competitive season of gameplay soccer heading.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Active player on the university's current team roster for the upcoming competitive season.
* Is eligible to participate in games and is not redshirting.

Exclusion Criteria:

* Is recovering from a Physician diagnosed concussion.
* Is recovering from another injury prohibiting the study participant from participating in all sport-related activities.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Collegiate women soccer players who actively compete at the NCAA Division 1-A competition level.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2023-11-09 (Actual)

PRIMARY OUTCOMES:
Change in plasma neurofilament light concentrations from baseline, during, and after a competitive season. | Baseline, 1 Months, 2 Months, 3 Months, 6 Months
  Plasma neurofilament light (pg/mL) is a biomarker of axonal brain injury following sports-related head impacts.
Change in purposeful soccer heading frequencies from baseline, during, and after a competitive season. | Baseline, 2 weeks, 4 weeks, 6 weeks, 8 weeks, 10 weeks, 12 weeks, 14 weeks
  HeadCount is a web-based, structured, self-administered questionnaire to assess longer-term heading frequencies (#) during competitive play and is administered bi-weekly.
Change in Omega-3 status from baseline, during, and after a competitive season. | Baseline, 1 Months, 2 Months, 3 Months, 6 Months
  Omega-3 Index (%) is the omega-3 fatty acid content of eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) within membrane of red blood cell. It is expressed as EPA+DHA as a percent of total identified fatty acids.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron F Carbuhn, PhD, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - University of Missouri Kansas City, Kansas City, Missouri
  - Rockhurst University, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: No